CLINICAL TRIAL: NCT04400071
Title: Biologic Mechanisms and Dosing of Active Music Engagement in Children With Acute Lymphoblastic Leukemia and Parents
Brief Title: Biology and Benefits of Music Play and Stories for Kids/Parents During ALL Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Children's Mercy Hospital Kansas City (Other); Ann & Robert H Lurie Children's Hospital of Chicago (Other); National Institute of Nursing Research (NINR) (NIH); James Whitcomb Riley Hospital for Children (Other); UCSF Benioff Children's Hospital Oakland (Other)
Responsible Party: Principal Investigator, Sheri Robb, Assistant Professor, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: R01NR019190 (NIH); 5R01NR019190-05 (NIH)
Record Dates: First submitted 2020-05-15; First posted 2020-05-22 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Acute Lymphoblastic Leukemia, Pediatric; Pediatric Cancer
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Study personnel responsible for administering self report measures will be blinded to participant's study condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Music Engagement (Experimental): See intervention description.
  Interventions: Behavioral: Active Music Engagement
- Audio Storybooks (Active Comparator): See intervention description.
  Interventions: Behavioral: Audio Storybooks

INTERVENTIONS:
Behavioral: Active Music Engagement — Weekly 45-minute sessions with a board-certified music therapist delivered during weekly clinic visits for the consolidation phase of ALL treatment. Children with standard risk ALL will receive 4 sessions over 4 weeks. Children with high risk ALL will receive 8 sessions over 8 weeks. Sessions are delivered in a private setting during regularly scheduled clinic appointments. During the first visit, parent and child will receive information on how they can use music play activities to help manage distress during treatment. The music therapist will lead parent and child in a variety of music play activities. Parent and child will receive a music kit that includes items such as hand-held rhythm instruments, puppets, and a music CD. During subsequent visits the music therapist will lead parent and child through the music play activities, answer questions, and make suggestions for using these activities in the hospital and at home.
  Arms: Active Music Engagement
Behavioral: Audio Storybooks — Weekly 45-minute sessions with a trained provider delivered during weekly clinic visits for the consolidation phase of ALL treatment. Children with standard risk ALL will receive 4 sessions over 4 weeks. Children with high risk ALL will receive 8 sessions over 8 weeks. Sessions are delivered in a private setting during regularly scheduled clinic appointments. Each session children/parents will choose and listen to one of three illustrated children's books with audio-recorded narration.
  Arms: Audio Storybooks

SUMMARY:
Music therapy has become a standard palliative care service in many pediatric and adult hospitals; however, a majority of music therapy research has focused on the use of music to improve psychosocial dimensions of health, without considering biological dimensions. This study builds on prior work examining the psychosocial mechanisms of action underlying an Active Music Engagement (AME) intervention, designed to help manage emotional distress and improve positive health outcomes in young children with cancer and parents, by examining its effects on biomarkers of stress and immune function. The purposes of this two group, randomized controlled trial are to examine biological mechanisms of effect and dose-response relationships of AME on child/parent stress during the consolidation phase of Acute Lymphoblastic Leukemia (ALL) treatment. Specific aims are to: Aim 1. Establish whether AME lowers child and parent cortisol during ALL treatment. Aim 2. Examine cortisol as a mediator of AME effects on child and parent outcomes during ALL treatment. Aim 3 (exploratory). Examine the dose-response relationship of AME on child and parent cortisol during ALL treatment. Findings will provide a more holistic understanding about how active music interventions work to mitigate cancer-related stress and its potential to improve immune function, with direct implications for the evidence-based use of music to improve health.

DETAILED DESCRIPTION:
Music therapy has become a standard palliative care service in many pediatric and adult hospitals. However, a majority of music therapy research has focused on the use of music to improve psychosocial dimensions of health, without considering biological dimensions. In addition, few studies have examined dose-response relationships. Cancer treatment is an inherently stressful experience, and a significant number of young children and parents (caregivers) experience persistent, interrelated emotional distress and poor quality of life. Many parents also experience traumatic stress symptoms because of their child's cancer diagnosis and treatment. The investigators previously tested an Active Music Engagement (AME) intervention that uses active music play to diminish stressful attributes of cancer treatment to help manage emotional/traumatic distress experienced by young children (ages 3-8) and parents and improve quality of life. A recent AME trial is examining psychosocial mechanisms of action responsible for change in child/parent outcomes. The current study expands on this work by examining AME's effects on several biomarkers to provide a more holistic understanding about how active music interventions work to mitigate cancer-related stress and its potential to improve immune function. The purposes of this two group, randomized controlled trial are to examine biological mechanisms of effect and dose-response relationships of AME on child/parent stress during the consolidation phase of Acute Lymphoblastic Leukemia (ALL) treatment. Specific aims are to: 1) establish whether AME lowers child and parent cortisol, 2) examine cortisol as a mediator of AME effects on child and parent outcomes, and 3) examine the dose-response relationship of AME on child and parent cortisol. Child/parent dyads (n=250) will be stratified (by age, site, ALL risk level) and randomized in blocks of four to AME or attention control. Each group will receive one 45-minute session during weekly clinic visits for the duration of ALL consolidation (4 weeks standard risk; 8 weeks high risk). Parents will complete measures at baseline and following the last study session. Child and parent salivary cortisol samples will be taken pre and post-session for the first 4 AME or attention control sessions. Child blood samples will be reserved from routine blood draws prior to sessions 1 and 4 (all participants) and session 8 (high risk participants). Linear mixed models will be used to estimate AME's effect on child and parent cortisol. Examining child and parent cortisol as mediators of AME effects on child and parent outcomes will be performed in an ANCOVA setting, fitting the appropriate mediation models using MPlus and then testing indirect effects using the percentile bootstrap approach to estimate the indirect effect. Graphical plots and non-linear repeated measures models will be used to examine the dose-response relationship of AME on child and parent cortisol.

ELIGIBILITY:
Inclusion Criteria:

* Child is 3 - 8 years of age at time of enrollment
* Child has diagnosis of standard or high risk B- or T-cell acute lymphoblastic leukemia (ALL) or lymphoblastic lymphoma (LyLy)
* Child is currently receiving induction therapy
* One parent (>18 years of age) can be present for all sessions.

Exclusion Criteria:

* Child has Ph+ ALL,
* Child has Cushing disease,
* Child is taking steroid medication for asthma and/or has asthma that is not well controlled,
* The parent does not speak English, or
* The child has a significant cognitive impairment that might hinder participation (determination made in consultation with attending physician, oncologist, and parents).

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 192 (Actual)
Dates: Start 2020-08-07 (Actual); Primary Completion 2025-04-11 (Actual); Study Completion 2025-04-11 (Actual)

PRIMARY OUTCOMES:
Change in Child and Parent Stress (Salivary Cortisol) | Pre/Post-Sessions 1, 2, 3, and 4 (each session is 7 days apart; each session has a 45 min. duration).
  We will measure salivary cortisol (a steroid hormone) as a biological indicator of stress. Cortisol is one of the most frequently used biomarkers for stress and has been used in several cancer studies.
Change in Immunomodulatory Cytokines (children only) (blood) | Pre-Session Week 1 and Week 4 (all child participants); and Pre-Session Week 8 (only high risk child participants).
  We will measure serum levels of IL-1β, IL-6, TNF-α, IFN-γ, IL-4, IL-10, and IL-13. The activation of the HPA-axis has been reported to shift to promote the secretion of anti-inflammatory cytokines (IL-4, IL-10, IL-13) and decrease pro-inflammatory cytokines (IL-1β, IL-6, TNF-α, IFN-γ) and thus modulate immune function.
Change in Child Health Questionnaire-Mental Health Subscale (CHQ) | Baseline; Post-Session Week 4 (standard risk participants); Post-Session Week 8 (high risk participants)
  Measures the frequency of both negative and positive states. Items capture anxiety, depression, and positive affect. We chose the parent-report version due to our targeted child age range of 3-8 years; parent-proxy and child self-report measures are scored differently, so we elected to use parent-proxy for all children. The subscale includes 16 parent-report items on a 5-point Likert-scale, ranging from 1 (none of the time) to 5 (all of the time). Scores range from 16-80 with higher scores indicating better mental health. Across 25 subgroups, the median Cronbach alpha coefficient for the subscale was .76, coefficients ranged from .67 to .86.
Change in KINDLR Questionnaire for Measuring Health-Related Quality of Life in Children | Baseline; Post-Session Week 4 (standard risk participants); Post-Session Week 8 (high risk participants).
  Measures global quality of life. The KINDL is used widely and has been translated into 11 languages. It was selected over other well-known measures for its positive health perspective, especially for younger children. The KINDL consists of 24 parent-report items rated on a 5-point Likert-scale, ranging from 1 (never) to 5 (all the time). There are 6 subscales: Physical well-being, Emotional Well-being, Self-Esteem, Family, Friends, and Everyday Functioning. We will use 20 items in 5 subscales, omitting the Everyday Functioning subscale, because it is focused on school-related functioning and children may not be attending school. Scores range from 20 - 100 with higher scores indicating better quality of life. KINDL parent-report is a valid and reliable measure for children as young as age 3. The KINDL has satisfactory convergent and discriminant validity, and a Cronbach alpha of .89 for the total scale.
Change in Profile of Mood States - Short Form (POMS-SF) | Baseline; Post-Session Week 4 (standard risk participants); Post-Session Week 8 (high risk participants).
  Measures mood disturbance. The scale is a self-report, 37-item instrument that yields scores on six subscales (tension-anxiety; depression-dejection; anger-hostility; vigor-activity; fatigue-inertia; confusion-bewilderment) and a total mood disturbance score. Respondents are given 37 adjectives used to describe feelings during the last week and asked to respond to each item using a 5-point Likert scale (0 = not at all; 4 = extremely). Higher scores equal greater mood disturbance. Construct validity is widely supported. The POMS-SF strongly correlates with the original 65-item POMS (r = 0.99) and is one of the most commonly used measures for parent emotional distress in pediatric cancer research.
Change in Impact of Events Scale - Revised (IES-R) | Baseline; Post-Session Week 4 (standard risk participants); Post-Session Week 8 (high risk participants).
  A 22-item measure that measures traumatic stress symptoms in response to a traumatic event that is specified in the instructions. In our study, parents will respond to items in reference to their child's cancer treatment as the stressor. The scale includes three subscales: intrusion, avoidance, and hyperarousal. Parents respond to each item using a 5-point Likert scale (0 = not at all; 4 = extremely). Higher scores indicate greater traumatic stress symptoms. The IES-R has been used in studies of childhood cancer patients and their parents. Cronbach's alpha for Intrusion, Avoidance, and Hyperarousal scales were .91, .84, and .90 respectively.
Change in Index of Well-being | Baseline; Post-Session Week 4 (standard risk participants); Post-Session Week 8 (high risk participants)
  A 9-item semantic differential scale describing present life using adjective extremes such as discouraging/hopeful. Higher scores mean greater well-being. The scale has well established construct validity and a reported Cronbach alpha of .93 for the total scale.

CONTACTS AND LOCATIONS:
Overall Officials: Sheri L Robb, PhD, Principal Investigator — Indiana University
Locations (4):
- United States (4):
  - UCSF Benioff Children's Hospital, Oakland, California
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Children's Mercy Hospital, Kansas City, Missouri

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Robb SL, Clair AA, Watanabe M, Monahan PO, Azzouz F, Stouffer JW, Ebberts A, Darsie E, Whitmer C, Walker J, Nelson K, Hanson-Abromeit D, Lane D, Hannan A. A non-randomized [corrected] controlled trial of the active music engagement (AME) intervention on children with cancer. Psychooncology. 2008 Jul;17(7):699-708. doi: 10.1002/pon.1301. PMID 18033724
- [Background] Robb SL, Haase JE, Perkins SM, Haut PR, Henley AK, Knafl KA, Tong Y. Pilot Randomized Trial of Active Music Engagement Intervention Parent Delivery for Young Children With Cancer. J Pediatr Psychol. 2017 Mar 1;42(2):208-219. doi: 10.1093/jpepsy/jsw050. PMID 27289068
- [Background] Robb SL. The effect of therapeutic music interventions on the behavior of hospitalized children in isolation: developing a contextual support model of music therapy. J Music Ther. 2000 Summer;37(2):118-46. doi: 10.1093/jmt/37.2.118. PMID 10932125
- [Derived] Robb SL, Russ KA, Holochwost SJ, Stegenga K, Perkins SM, Jacob SA, Henley AK, MacLean JA. Protocol and biomarker strategy for a multi-site randomized controlled trial examining biological mechanisms and dosing of active music engagement in children with acute lymphoblastic leukemia and lymphoma and parents. BMC Complement Med Ther. 2023 Mar 27;23(1):90. doi: 10.1186/s12906-023-03909-w. PMID 36973774